CLINICAL TRIAL: NCT00006039
Title: Phase II Study of Weekly Administered High-Dose Pegylated Interferon Alfa-2B (PEGIntron) in Advanced Stage Low Grade Non-Hodgkin's Lymphoma
Brief Title: Interferon Alfa-2b in Treating Patients With Advanced Low-Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-101; CDR0000068054 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1814
Record Dates: First submitted 2000-07-05; First posted 2004-05-03 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma; Small Intestine Cancer
Keywords: small intestine lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell

INTERVENTIONS:
Biological: pegylated interferon alfa

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of the cancer cells and slow the growth of non-Hodgkin's lymphoma.

PURPOSE: Phase II trial to study the effectiveness of interferon alfa-2b in treating patients who have advanced low-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response in patients with minimally treated or previously untreated advanced low-grade non-Hodgkin's lymphoma treated with pegylated interferon alfa-2b. II. Determine the effects of this treatment regimen on the immune system by measuring T-cell subsets and NK cells in this patient population. III. Determine event-free and progression-free survival in this patient population treated with this regimen. IV. Evaluate the toxicity profile of this treatment regimen in these patients.

OUTLINE: Patients receive pegylated interferon alfa-2b subcutaneously once weekly for 6 months in the absence of disease progression or unacceptable toxicity. Upon completion of treatment, patients are followed every 6 months for at least 2 years.

PROJECTED ACCRUAL: A total of 30 patients will be initially accrued for this study. Additional patients will be accrued if acceptable responses are seen in the first cohort.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed low-grade lymphoma including any of the following: REAL classification Follicular lymphoma (grade I or II) Lymphoplasmacytoid lymphoma Small lymphocytic lymphoma Marginal B-cell lymphoma MALT lymphoma International Working Formulation Follicular small cleaved cell lymphoma Follicular mixed small and large cell lymphoma Small lymphocytic lymphoma No intermediate or high-grade non-Hodgkin's lymphoma (NHL) histology No evidence of histologic transformation If previously untreated, large tumor burden including any of the following: Nodal or extranodal mass greater than 7 cm in diameter Involvement of at least 3 nodal sites (each greater than 3 cm in diameter) Systemic symptoms Splenomegaly Ureteral compression Intraabdominal stage II, stage III, or stage IV disease Measurable disease No prior systemic therapy OR No more than 1 prior therapy ( e.g., chemotherapy, immunotherapy, chemotherapy with immunotherapy, or chemotherapy with regional radiotherapy) A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC greater than 2,000/mm3 Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 75,000/mm3 Hemoglobin greater than 10 g/dL Absolute lymphocyte count no greater than 5,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) SGOT/SGPT less than 2.5 times ULN Alkaline phosphatase less than 2.5 times ULN No active hepatitis Renal: Creatinine less than 1.5 times ULN OR Creatinine clearance greater than 60 mL/min Cardiovascular: No severe cardiovascular disease No myocardial infarction within the past 6 months No unstable angina No class III or IV congestive heart failure No ventricular tachyarrhythmias Other: No active uncontrolled infections or infections requiring systemic antibiotics HIV negative No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix No history of neuropsychiatric disorder requiring hospitalization Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 12 weeks since prior immunotherapy (e.g., rituximab) No prior cytokines (except filgrastim (G-CSF) or epoetin alfa) Chemotherapy: See Disease Characteristics Endocrine therapy: No concurrent systemic corticosteroids Radiotherapy: See Disease Characteristics Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol S. Portlock, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States